CLINICAL TRIAL: NCT01264588
Title: A Randomized, Single Blind, Comparative, Controlled Study On The Effects Of Topical Calcium Glycerophosphate On Surgical Wound Healing And Residual Scarring In Bilateral Total Knee Arthroplasty Patients
Brief Title: The Effects of Topical Calcium Glycerophosphate on Surgical Wound Healing and Residual Scarring
Acronym: TOPCGP-2008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AkPharma Inc. (Industry)
Collaborators: Rothman Institute Orthopaedics (Other); Texas Tech University Health Sciences Center (Other); Cyberderm Inc. (Industry); Bacharach Institute for Rehabilitation, Pomona, NJ (Other)
Responsible Party: Alvin C. Ong, M.D., Rothman Institute Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TOPCGP-2008
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Wound Healing; Scarring
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- topical calcium glycerophosphate lotion (Active Comparator)
  Interventions: Other: Topical calcium glycerophosphate lotion
- standard-of-care (No Intervention)

INTERVENTIONS:
Other: Topical calcium glycerophosphate lotion — 2g once daily for 6 weeks (post-op day 3 thru 42)
  Arms: topical calcium glycerophosphate lotion

SUMMARY:
The purpose of this study is to determine whether topical application of calcium glycerophosphate will result in superior wound appearance and scar minimization.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained
* 45-75 years of age
* Scheduled for bilateral knee replacement surgery

Exclusion Criteria:

* Employee or immediate family of either AkPharma or employee or immediate family of investigator or site personnel
* Pregnant or breast feeding Known allergy or hypersensitivity to calcium or phosphorus supplements
* Diagnosed with type I or type II diabetes mellitus

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Improvement of surgical wound appearance | Post-Op Day: 3 (baseline), 7, 14, 42, 70, 98, 180, 365
  Digital photographs as objective measurements are taken at each time point, and evaluated by an Expert Grader, blinded as to treatment vs. control, for any differences in the time required for wound closure and/ or scar minimization between treated and untreated groups.

SECONDARY OUTCOMES:
Reduction of visible erythema/ inflammation | Post-Op Day: 3 (baseline), 7, 14, 42, 70, 98, 180, 365
  Digital photographs as objective measurements are taken at each time point, and evaluated by an Expert Grader, blinded as to treatment vs. control, for any differences in reduction of visible erythema/ inflammation between treated and untreated groups.
Scar minimization or prevention | Post-Op Day: 3 (baseline), 7, 14, 42, 70, 98, 180, 365
  Digital photographs as objective measurements are taken at each time point, and evaluated by an Expert Grader, blinded as to treatment vs. control, for any differences in scar appearance between treated and untreated groups.
Incision/ scar pain and sensitivity | Post-Op Day: 3 (baseline), 7, 14, 42, 70, 98, 180, 365
  Subjects are asked to rate their pain at the site of incision for each knee, using a scale of 0 (no pain) to 10 (excruciating pain). The pain evaluations are recorded on a pain diary sheet provided at each time point.
Range of motion | Post-Op Day: 3 (baseline), 7, 42, 180, 365
  Range of motion (both flexion and extension) is evaluated using standard goniometric methods.

CONTACTS AND LOCATIONS:
Overall Officials: Alvin C. Ong, M.D., Principal Investigator — Rothman Institute Orthopaedics
Locations (1):
- Rothman Institute Orthopaedics, Egg Harbor, New Jersey, United States